CLINICAL TRIAL: NCT00655590
Title: A Randomized, Double-blind, Placebo Controlled, Parallel Arm, Multicenter Trial Assessing the Effect of Daily Treatment of Vardenafil 20 mg or Sildenafil 100 mg Compared to Placebo on Spermatogenesis
Brief Title: Assess the Effect of Daily Treatment of Vardenafil 20mg or Sildenafil 100mg and Placebo on Sperm Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11520
Record Dates: First submitted 2008-04-04; First posted 2008-04-10 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction; Sildenafil; Vardenafil; Spermatogenesis; Sperm concentration; Sperm count; Morphology; Motility; Reproductive hormonal
MeSH Terms: conditions — Erectile Dysfunction | interventions — Vardenafil Dihydrochloride; Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Drug: Levitra (Vardenafil, BAY38-9456)
- Arm 2 (Active Comparator)
  Interventions: Drug: Sildenafil
- Arm 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levitra (Vardenafil, BAY38-9456) — 20 mg daily dosing
  Arms: Arm 1
Drug: Sildenafil — 100 mg daily dosing
  Arms: Arm 2
Drug: Placebo — Matching placebos
  Arms: Arm 3

SUMMARY:
Assess the effect of daily treatment of vardenafil 20mg or sildenafil 100mg and placebo on sperm function

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects or men with ED aged 25 - 64
* Baseline sperm conc. of > 20 mio / ml- Normal World Health Organization A+B+C sperm mortality > 50%- Normal sperm morphology (WHO, 1992 manual criteria) > 30% and - 1.0 mL ejaculate volume at each of the 3 analyses during the screening phase.

Exclusion Criteria:

* Presence of any psychological or physiological abnormalities that in the opinion of the Investigator would significantly impair sexual performance or ability to provide semen samples according to the protocol- Spinal cord injury
* History of surgical prostatectomy
* Other exclusion criteria apply according to US Product Information

Ages: 25 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2005-01; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Proportion of vardenafil subjects with a 50% or greater decrease from baseline in mean sperm concentration at 6 months (LOCF), compared to placebo after repeated use | 24 weeks

SECONDARY OUTCOMES:
Mean sperm concentration | 24 weeks
Mean sperm count | 24 weeks
Sperm morphology | 24 weeks
Sperm motility | 24 weeks
Reproductive hormones | 24 weeks
Proportion of sildenafil subjects with a 50% or greater decrease from baseline in mean sperm concentration at 6 months (LOCF), compared to placebo and vardenafil after repeated use | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (18):
- United States (18):
  - Phoenix, Arizona
  - Tempe, Arizona
  - Beverly Hills, California
  - La Mesa, California
  - Laguna Hills, California
  - San Diego, California
  - Torrance, California
  - Van Nuys, California
  - Waterbury, Connecticut
  - Aventura, Florida
  - New Orleans, Louisiana
  - Ann Arbor, Michigan
  - Minneapolis, Minnesota
  - Rochester, Minnesota
  - Great Neck, New York
  - New York, New York
  - Cincinnati, Ohio
  - San Antonio, Texas